CLINICAL TRIAL: NCT06339801
Title: Role of Mucosal Impedance Measurement for the Diagnosis of Gastroesophageal Reflux Disease
Status: Recruiting | Type: Observational
Sponsor: Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Maria Marta Piskorz, Principal Investigator, Hospital de Clinicas José de San Martín
Other Study IDs: HCJSM-24-193
Record Dates: First submitted 2024-03-19; First posted 2024-04-01 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Gastroesophageal Reflux
Keywords: gastroesophageal reflux; mucosal impedance
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- GERD group: Patients >18 years presenting symptoms of GERD that have not adequately responded to proton pump inhibitors (PPIs) treatment after 8 weeks and have undergone upper gastrointestinal endoscopy (UGIE) without erosive esophagitis.
  Patients with a broad spectrum of severity, assessed through the GERDq score, will be included
  Interventions: Device: MiVu

INTERVENTIONS:
Device: MiVu — All patients will undergo mucosal impedance (MI) measurement using the MiVu™ Mucosal Integrity Testing System (Diversatek Healthcare, Inc.).

SUMMARY:
Existing current tests for diagnosing GERD are suboptimal because they lack adequate sensitivity or specificity. Upper gastrointestinal endoscopy is highly specific for diagnosing GERD, particularly when erosive esophagitis is present (Los Angeles Classification B, C, or D). Nevertheless, its sensitivity is limited, as this scenario is only present in 30% of cases. Most patients will exhibit normal endoscopic findings, indicating Non-Erosive Reflux Disease (NERD). The 24-hour impedance-pH monitoring (MII) is currently considered the gold standard. However, its main limitation is that it can only measure reflux activity over a 24-hour period, in addition to the discomfort caused by the catheter. 6-8 It is noteworthy that 50% of patients with NERD will have pathological reflux, and the other 50% will have a sensory disorder. The importance of making an accurate diagnosis lies in the treatment, which varies in each case.11 Recently, a minimally invasive device was developed and validated in the USA to assess changes in esophageal mucosal impedance. This serves as a tool for evaluating tissue changes associated with chronic reflux. However, this device has recently undergone improvements. This new technology has not been tested yet for GERD diagnosis. The primary benefit would be the ability to diagnose GERD in symptomatic patients with NERD during the initial endoscopy conducted under sedation.

Objectives

The Main objectives of this study are to:

1. Evaluate the diagnostic performance of mucosal impedance measurement.
2. Investigate the mucosal impedance pattern in patients with and without GERD.

Secondary objectives:

1. Evaluate the correlation between the global mucosal impedance measurement vs the first 3cm measurement
2. Evaluate the best probability score to distinguish between GERD and non-GERD Design Prospective, cross-sectional, and analytical study Study Design and Procedures The study will be conducted in the Gastroenterology Department of the Hospital de Clínicas José de San Martin, University of Buenos Aires, Argentina. Following a 4-week screening period during which a proton pump inhibitor (PPI) washout will be performed, and baseline measurements will be taken, all patients will undergo upper gastrointestinal endoscopy with mucosal impedance measurement and 24-hour impedance/pH monitoring.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease (GERD) occurs when gastroduodenal content refluxes, causing bothersome symptoms and/or complications. 1 It is estimated that GERD affects 20-30% of the population in Western countries 2 (23% in Argentina), and it is associated with an impairment in the quality of life and significant healthcare costs. 3-5 Existing current tests for diagnosing GERD are suboptimal because they lack adequate sensitivity or specificity. Upper gastrointestinal endoscopy is highly specific for diagnosing GERD, particularly when erosive esophagitis is present (Los Angeles Classification B, C, or D). Nevertheless, its sensitivity is limited, as this scenario is only present in 30% of cases. Most patients will exhibit normal endoscopic findings, indicating Non-Erosive Reflux Disease (NERD). The 24-hour impedance-pH monitoring (MII) is currently considered the gold standard. However, its main limitation is that it can only measure reflux activity over a 24-hour period, in addition to the discomfort caused by the catheter. 6-8 The last Lyon Consensus considered GERD when erosive esophagitis is present (Los Angeles Classification B, C, or D) or acid exposure time (AET) is >6% on ambulatory studies. Acid exposure time <4% definitively rules out pathologic gastroesophageal acid reflux, while AET between 4-6% is considered borderline. 9,10 It is noteworthy that 50% of patients with NERD will have pathological reflux, and the other 50% will have a sensory disorder. The importance of making an accurate diagnosis lies in the treatment, which varies in each case.11 Recently, a minimally invasive device was developed and validated in the USA to assess changes in esophageal mucosal impedance. This serves as a tool for evaluating tissue changes associated with chronic reflux.12 However, this device has recently undergone improvements. This new technology has not been tested yet for GERD diagnosis. The primary benefit would be the ability to diagnose GERD in symptomatic patients with NERD during the initial endoscopy conducted under sedation.

Objectives

The Main objectives of this study are to:

1. Evaluate the diagnostic performance of mucosal impedance measurement.
2. Investigate the mucosal impedance pattern in patients with and without GERD.

Secondary objectives:

1. Evaluate the correlation between the global mucosal impedance measurement vs the first 3cm measurement
2. Evaluate the best probability score to distinguish between GERD and non-GERD Design Prospective, cross-sectional, and analytical study METHODS Participants, Interventions, and Outcomes. Study Setting Inclusion Criteria Patients >18 years presenting symptoms of GERD that have not adequately responded to proton pump inhibitors (PPIs) treatment after 8 weeks and have undergone upper gastrointestinal endoscopy (UGIE) without erosive esophagitis.

Patients with a broad spectrum of severity, assessed through the GERDq score, will be included Exclusion Criteria

* Pregnancy or lactation
* Esophageal disorders (esophageal motor disorders, eosinophilic esophagitis, neoplastic diseases)
* Uncontrolled systemic diseases (diabetes mellitus, hypo- or hyperthyroidism, cancer, etc.)
* Lack of informed consent
* Severe psychiatric disorders Study Design and Procedures The study will be conducted in the Gastroenterology Department of the Hospital de Clínicas José de San Martin, University of Buenos Aires, Argentina. Following a 4-week screening period during which a proton pump inhibitor (PPI) washout will be performed, and baseline measurements will be taken, all patients will undergo upper gastrointestinal endoscopy with mucosal impedance measurement and 24-hour impedance/pH monitoring.

Intervention All patients will undergo mucosal impedance (MI) measurement using the MiVu™ Mucosal Integrity Testing System (Diversatek Healthcare, Inc.). The MiVu™ Mucosal Integrity Testing System utilizes a device (MiVu™ Endo Cap) that attaches to the distal end of the endoscope, along with proprietary software to instantly detect changes in esophageal mucosal integrity during endoscopy. Patients are required to fast for 8 hours before the procedure. During an upper gastrointestinal endoscopy under anesthesia sedation, measurements are taken from direct contact of the sensors with the esophageal mucosa. Any luminal air or liquid between the sensors and mucosal tissue will be pressed away from the tissue being measured. After identifying the gastroesophageal junction, measurements will be initiated 2cm above it. The endoscopist will wait until all 3 sensors make stable contact with the mucosa, indicated by high-quality signals marked in green color by the software. The Study Metrics require data spanning 10 consecutive centimeters. Each measurement capture will span 3 cm, and a minimum of 4 measurements spanning 10 cm are required. Once measurements have been captured at 4 depths, the metrics will populate. MI measurements will be expressed in Ohms and analyzed using the ZVU software version 3.3 or greater (Diversatek Healthcare, Inc.). Once 10 centimeters worth of consecutive data have been acquired, the probabilities of disease will be displayed and patients will be categorized as: 1) NERD and 2) Non-NERD based on the measurement result. The results will be expressed in Ohms, and the interpretation will be based on the results from table 2 in the previous MI validation publication.14 Subsequently, a 24-hour impedance/pH monitoring without proton pump inhibitors (PPI), preceded by high-resolution esophageal manometry to identify the lower esophageal sphincter height, will be performed. Both assessments will be conducted by different operators in a blind and independent manner.

Patients will be divided into two groups: A) NERD: when the percentage of time of acid exposure is greater than 6%, B) Non-NERD: when the percentage of acid exposure is less than 4%. The Demeester score will be reported for both groups.

Treatment response evaluation

Based on the previously described categorization, the following treatment will be initiated:

1. Dexlansoprazole 30mg per day in the GERD group
2. Amitriptyline 10mg per day in the non-GERD group At 8 weeks post-treatment, a GerdQ assessment will be conducted. Sample Size Considering an estimated sensitivity of mucosal impedance measurement for the diagnosis of GERD of 70%, a sample size of 100 patients was calculated. Factoring in a 20% patient loss, a total of 120 patients will be screened.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years presenting symptoms of GERD that have not adequately responded to proton pump inhibitors (PPIs) treatment after 8 weeks and have undergone upper gastrointestinal endoscopy (UGIE) without erosive esophagitis.

Patients with a broad spectrum of severity, assessed through the GERDq score, will be included

Exclusion Criteria:

* ● Pregnancy or lactation

  * Esophageal disorders (esophageal motor disorders, eosinophilic esophagitis, neoplastic diseases)
  * Uncontrolled systemic diseases (diabetes mellitus, hypo- or hyperthyroidism, cancer, etc.)
  * Lack of informed consent
  * Severe psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years presenting symptoms of GERD that have not adequately responded to proton pump inhibitors (PPIs) treatment after 8 weeks and have undergone upper gastrointestinal endoscopy (UGIE) without erosive esophagitis.
  Patients with a broad spectrum of severity, assessed through the GERDq score, will be included
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
diagnostic performance | immediately after the intervention/procedure
  diagnostic performance of mucosal impedance measurement
mucosal impedance pattern | immediately after the intervention/procedure
  mucosal impedance pattern in patients with and without GERD.

SECONDARY OUTCOMES:
Correlations | immediately after the intervention/procedure
  correlation between the global mucosal impedance measurement vs the first 3cm measurement
Probability score | immediately after the intervention/procedure
  the best probability score to distinguish between GERD and non-GERD

CONTACTS AND LOCATIONS:
Overall Officials: JORGE A OLMOS, MD, Principal Investigator — HOSPITAL DE CLINICAS JOSE DE SAN MARTIN
Locations (1):
- Hospital de Clinicas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martinez SD, Malagon IB, Garewal HS, Cui H, Fass R. Non-erosive reflux disease (NERD)--acid reflux and symptom patterns. Aliment Pharmacol Ther. 2003 Feb 15;17(4):537-45. doi: 10.1046/j.1365-2036.2003.01423.x. PMID 12622762
- [Background] Gyawali CP, Yadlapati R, Fass R, Katzka D, Pandolfino J, Savarino E, Sifrim D, Spechler S, Zerbib F, Fox MR, Bhatia S, de Bortoli N, Cho YK, Cisternas D, Chen CL, Cock C, Hani A, Remes Troche JM, Xiao Y, Vaezi MF, Roman S. Updates to the modern diagnosis of GERD: Lyon consensus 2.0. Gut. 2024 Jan 5;73(2):361-371. doi: 10.1136/gutjnl-2023-330616. PMID 37734911